CLINICAL TRIAL: NCT00907985
Title: Double Blind, Double-dummy, Randomised, Placebo Controlled Study to Evaluate the Effect of Single Doses of Drug A (Lamotrigine) and Drug B (Vofopitant) Alone and in Combination on Resting Motor Threshold in Healthy Subjects
Brief Title: A Study to Evaluate the Effect of Single Doses of Drug A (Lamotrigine) and Drug B (Vofopitant) Alone and in Combination on Resting Motor Threshold in Healthy Subjects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow recruitment; trial unlikely to reach completion
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 112676
Record Dates: First submitted 2009-05-07; First posted 2009-05-25 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Bipolar Disorder
Keywords: Healthy Volunteer; Resting motor threshold (rMT); Transcranial magnetic stimulation (TMS)
MeSH Terms: conditions — Bipolar Disorder | interventions — vofopitant; Lamotrigine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (20):
- Treatment sequence A (Experimental): Subjects on sequence A will receive single dose of vofopitant 10 milligrams capsule in part 1, single doses of lamotrigine 175 milligrams tablet + vofopitant 10 milligrams capsule in session A of part 2 and placebo + vofopitant 10 milligrams capsule in session B of part 2.
  Interventions: Drug: Placebo; Drug: Vofopitant; Drug: Lamotrigine
- Treatment sequence B (Experimental): Subjects on sequence B will receive single dose of vofopitant 10 milligrams capsule in part 1, single doses of placebo + vofopitant 10 milligrams capsule in session A of part 2 and lamotrigine 175 milligrams tablet + vofopitant 10 milligrams capsule in session B of part 2.
  Interventions: Drug: Placebo; Drug: Vofopitant; Drug: Lamotrigine
- Treatment sequence C (Experimental): Subjects on sequence C will receive single dose of placebo in part 1, single doses of lamotrigine 175 milligrams tablet + vofopitant 10 milligrams capsule in session A of part 2 and placebo + vofopitant 10 milligrams capsule in session B of part 2.
  Interventions: Drug: Placebo; Drug: Vofopitant; Drug: Lamotrigine
- Treatment sequence D (Experimental): Subjects on sequence D will receive single dose of placebo in part 1, single doses of placebo + vofopitant 10 milligrams capsule in session A of part 2 and lamotrigine 175 milligrams tablet + vofopitant 10 milligrams capsule in session B of part 2.
  Interventions: Drug: Placebo; Drug: Vofopitant; Drug: Lamotrigine
- Treatment sequence E (Experimental): Subjects on sequence E will receive single dose of vofopitant 10 milligrams capsule in part 1, single doses of lamotrigine 175 milligrams tablet + vofopitant 10 milligrams capsule in session A of part 2 and placebo + placebo in session B of part 2.
  Interventions: Drug: Placebo; Drug: Vofopitant; Drug: Lamotrigine
- Treatment sequence F (Experimental): Subjects on sequence F will receive single dose of vofopitant 10 milligrams capsule in part 1, single doses of placebo + placebo in session A of part 2 and lamotrigine 175 milligrams tablet + vofopitant 10 milligrams capsule in session B of part 2.
  Interventions: Drug: Placebo; Drug: Vofopitant; Drug: Lamotrigine
- Treatment sequence G (Experimental): Subjects on sequence G will receive single dose of placebo in part 1, single doses of lamotrigine 175 milligrams tablet + vofopitant 10 milligrams capsule in session A of part 2 and placebo + placebo in session B of part 2.
  Interventions: Drug: Placebo; Drug: Vofopitant; Drug: Lamotrigine
- Treatment sequence H (Experimental): Subjects on sequence H will receive single dose of placebo part 1, single doses of placebo + placebo in session A of part 2 and lamotrigine 175 milligrams tablet + vofopitant 10 milligrams capsule in session B of part 2.
  Interventions: Drug: Placebo; Drug: Vofopitant; Drug: Lamotrigine
- Treatment sequence I (Experimental): Subjects on sequence I will receive single dose of vofopitant 10 milligrams capsule in part 1, single doses of lamotrigine 175 milligrams tablet + placebo in session A of part 2 and placebo + vofopitant 10 milligrams capsule in session B of part 2.
  Interventions: Drug: Placebo; Drug: Vofopitant; Drug: Lamotrigine
- Treatment sequence J (Experimental): Subjects on sequence J will receive single dose of vofopitant 10 milligrams capsule in part 1, single doses of placebo + vofopitant 10 milligrams capsule in session A of part 2 and lamotrigine 175 milligrams tablet + placebo in session B of part 2.
  Interventions: Drug: Placebo; Drug: Vofopitant; Drug: Lamotrigine
- Treatment sequence K (Experimental): Subjects on sequence K will receive single dose of placebo in part 1, single doses of lamotrigine 175 milligrams tablet + placebo in session A of part 2 and placebo + vofopitant 10 milligrams capsule in session B of part 2.
  Interventions: Drug: Placebo; Drug: Vofopitant; Drug: Lamotrigine
- Treatment sequence L (Experimental): Subjects on sequence L will receive single dose of placebo in part 1, single doses of placebo + vofopitant 10 milligrams capsule in session A of part 2 and lamotrigine 175 milligrams tablet + placebo in session B of part 2.
  Interventions: Drug: Placebo; Drug: Vofopitant; Drug: Lamotrigine
- Treatment sequence M (Experimental): Subjects on sequence M will receive single dose of vofopitant 10 milligrams capsule in part 1, single doses of lamotrigine 175 milligrams tablet + placebo in session A of part 2 and placebo + placebo in session B of part 2.
  Interventions: Drug: Placebo; Drug: Vofopitant; Drug: Lamotrigine
- Treatment sequence N (Experimental): Subjects on sequence N will receive single dose of vofopitant 10 milligrams capsule in part 1, placebo + placebo in session A of part 2 and lamotrigine 175 milligrams tablet + placebo in session B of part 2.
  Interventions: Drug: Placebo; Drug: Vofopitant; Drug: Lamotrigine
- Treatment sequence O (Experimental): Subjects on sequence O will receive placebo in part 1, single doses of lamotrigine 175 milligrams tablet + placebo in session A of part 2 and placebo + placebo in session B of part 2.
  Interventions: Drug: Placebo; Drug: Vofopitant; Drug: Lamotrigine
- Treatment sequence P (Experimental): Subjects on sequence P will receive placebo in part 1, single doses of placebo + placebo in session A of part 2 and lamotrigine 175 milligrams tablet + placebo in session B of part 2.
  Interventions: Drug: Placebo; Drug: Vofopitant; Drug: Lamotrigine
- Treatment sequence Q (Experimental): Subjects on sequence Q will receive single dose of vofopitant 10 milligrams capsule in part 1, single doses of lamotrigine 175 milligrams tablet + lamotrigine 150 milligrams tablet in session A of part 2 and placebo + placebo in session B of part 2.
  Interventions: Drug: Placebo; Drug: Vofopitant; Drug: Lamotrigine
- Treatment sequence R (Experimental): Subjects on sequence R will receive single dose of vofopitant 10 milligrams capsule in part 1, single doses of placebo + placebo in session A of part 2 and lamotrigine 175 milligrams tablet + lamotrigine 150 milligrams tablet in session B of part 2.
  Interventions: Drug: Placebo; Drug: Vofopitant; Drug: Lamotrigine
- Treatment sequence S (Experimental): Subjects on sequence S will receive placebo in part 1, single doses of lamotrigine 175 milligrams tablet + lamotrigine 150 milligrams tablet in session A of part 2 and placebo + placebo in session B of part 2.
  Interventions: Drug: Placebo; Drug: Vofopitant; Drug: Lamotrigine
- Treatment sequence T (Experimental): Subjects on sequence T will receive placebo in part 1, single doses of placebo + placebo in session A of part 2 and lamotrigine 175 milligrams tablet + lamotrigine 150 milligrams tablet in session B of part 2.
  Interventions: Drug: Placebo; Drug: Vofopitant; Drug: Lamotrigine

INTERVENTIONS:
Drug: Placebo — Single dose of placebo will be provided.
Drug: Vofopitant — Vofopitant (GR205171) will be provided as 5 milligram single dose capsule administered orally. It will be available as swedish orange, size 0 capsules.
Drug: Lamotrigine — Lamotrigine will be provided as 25 milligrams or 100 milligrams single dose dispersible tablet administered orally.

SUMMARY:
The purpose of this study is to investigate the effect of drug A on its own and when it is given in combination with drug B on markers of brain activity. The study will

1. Assess the effects of drug A and drug B on muscle movement after brain stimulation;
2. Examine how the body handles (absorbs, distributes, breaks down and gets rid of) drug A and drug B when given in combination;
3. Examine the safety of drug A and drug B when given together.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subject
* Male aged 18-65
* Greater than 50kg weight
* BMI 19-29.9 kg/m2

Exclusion Criteria:

* Positive drug/alcohol screen
* Positive HIV antibody
* History of drug dependence
* History of neurological disease
* Pacemaker
* Smoker

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-05-15 (Actual); Primary Completion 2010-06-10 (Actual); Study Completion 2010-06-10 (Actual)

PRIMARY OUTCOMES:
Effect of the study treatments on Resting Motor Thresholds (rMT) | Within 24 hours

SECONDARY OUTCOMES:
The safety and tolerability of the combination of study treatments. | Within 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Göttingen, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 112676 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/112676?search=study&study_ids=112676#rs
- Available data/document: Informed Consent Form: 112676 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 112676 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 112676 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 112676 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 112676 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 112676 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 112676 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register